CLINICAL TRIAL: NCT00229515
Title: Multicentre 2x2 Factorial Randomised Study Comparing Tirofiban Administered With the Single High-Dose Bolus Versus Abciximab and Sirolimus Eluting Stent Versus Bare Metal Stent in Acute Myocardial Infarction - MULTI-STRATEGY Trial
Brief Title: Multicentre 2x2 Factorial Randomised Study Comparing Tirofiban Versus Abciximab and SES Versus BMS in AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marco Valgimigli (Other)
Responsible Party: Sponsor-Investigator, Marco Valgimigli, Head of the Catheterization laboratory, Università degli Studi di Ferrara
Organization: Università degli Studi di Ferrara (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TSES-02-III
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Revascularization; Stent; ST segment elevation
MeSH Terms: conditions — Myocardial Infarction | interventions — Stents; Abciximab; Drug-Eluting Stents; Tirofiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Patients will receive abciximab infusion at standard regimen prior undergoing percutaneous coronary intervention for STEMI followed by BMS implantation in the culprit lesion
  Interventions: Other: abciximab followed by implantation of bare metal stent
- 2 (Experimental): Abciximab followed by implantation of sirolimus-eluting stent in the culprit lesion
  Interventions: Other: abciximab and Sirolimus eluting stent
- 3 (Experimental): tirofiban infusion followed by bare metal stent implantation
  Interventions: Other: tirofiban and bare metal stent
- 4 (Experimental): tirofiban and sirolimus-eluting stent
  Interventions: Other: tirofiban and sirolimus-eluting stent

INTERVENTIONS:
Other: abciximab followed by implantation of bare metal stent — Patients will receive infusion of abciximab at standard regimen before undergoing intervention for STEMI and then bare metal stent implantation in the culprit lesion
  Other Names: Glycoprotein IIB/IIIa inhibitors; Stent
  Arms: 1
Other: abciximab and Sirolimus eluting stent — Patients will receive abciximab infusion at standard regimen followed by implantation of sirolimus-eluting stent in the culprit lesion
  Other Names: glycoprotein IIb/IIIa inhibitors; stent; DES; drug-eluting stent
  Arms: 2
Other: tirofiban and bare metal stent — Patients will receive tirofiban infusion at high loading dose followed by standard infusion for 18-24 hours and subsequently they will be treated with bare metal stent implantation
  Other Names: glycoprotein IIb/IIIa inhibitors; stent; uncoated stent; bare metal stent
  Arms: 3
Other: tirofiban and sirolimus-eluting stent — Patients will receive tirofiban infusion at high loading dose followed by standard infusion for 18-24 hours and subsequently they will be treated with sirolimus-eluting stent implantation
  Other Names: glycoprotein IIb/IIIa inhibitors; stent; drug-eluting stent; sirolimus-eluting stent; DES; SES
  Arms: 4

SUMMARY:
The purpose of this study is to determine which from the four combinations tirofiban+sirolimus eluting stent (SES), tirofiban+bare metal stent (BMS), abciximab+SES, abciximab+BMS is the possible gold standard treatment for ST-segment elevation myocardial infarction in terms of efficacy and cost-efficacy.

DETAILED DESCRIPTION:
The combination abciximab plus bare metal stent (BMS) is currently considered the standard therapy for AMI. The use of sirolimus eluting stent (SES) is related to a reduction of the need for urgent target vessel revascularization (TVR). With current acquisition prices for abciximab and SES, replacing abciximab with tirofiban, administered as a single high-dose bolus (SHDB) regimen, is a promising strategy that would preserve financial resources. In a recent study the combination tirofiban and SES resulted to be associated to an overall lower major adverse cardiovascular events (MACE) rate with respect to the abciximab plus BMS. However, since no conclusion can be drawn yet regarding the relative contribution of a specific GP IIb/IIIa inhibitor or a stent type with respect to the other, the combination of abciximab and SES may be associated to an even lower event rate with respect to SHDB tirofiban and SES, thus offsetting the higher initial cost.

Comparison(s): four strategies (SHDB tirofiban + BMS, SHDB tirofiban + SES, abciximab + BMS, abciximab + SES) are compared to determine the possible gold standard treatment for ST-segment elevation myocardial infarction in terms of efficacy and cost-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* ST segment elevation myocardial infarction
* Schedule for primary percutaneous coronary intervention
* Informed consent

Exclusion Criteria:

* Administration of fibrinolytic or any GP IIb/IIIa inhibitors for the treatment of current acute myocardial infarction or within 1 month before it
* History of bleeding diathesis or allergy to the studies drug
* Major surgery within 30 days
* Limited life expectancy, e.g. neoplasms, others
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
The evaluation of the degree of ST-segment resolution after the mechanical intervention. | 90 minutes after last balloon inflation
The cumulative rate of death for any cause, reinfarction and target vessel revascularisation | 8 months

SECONDARY OUTCOMES:
Death, recurrent acute myocardial infarction, target vessel revascularization and target lesion revascularisation, considered separately or in combination. | at any time during follow-up
The evaluation of the cost-effectiveness of the involved experimental treatments. | 8 months, 1,3 and 5 years
stent thrombosis according to the ARC classification | any time during follow-up
the degree of cumulative or single lead ST segment resolution at time frames different from the primary endpoint. the degree of residual ST segment elevation. | immediately after intervention, at 90 minutes and at discharge
bleeding rate defined according to different classifications including TIMI, Acuity, GUSTO and Steeple. | at 30 days, 1 year, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Ferrari, Professor, Study Chair — Cattedra di Cardiologia, Azienda Ospedaliera Universitaria di Ferrara, Italy
Locations (1):
- Cattedra di Cardiologia, Azienda Ospedaliera Universitaria di Ferrara, Ferrara, Italy

REFERENCES:
- [Background] Valgimigli M, Percoco G, Malagutti P, Campo G, Ferrari F, Barbieri D, Cicchitelli G, McFadden EP, Merlini F, Ansani L, Guardigli G, Bettini A, Parrinello G, Boersma E, Ferrari R; STRATEGY Investigators. Tirofiban and sirolimus-eluting stent vs abciximab and bare-metal stent for acute myocardial infarction: a randomized trial. JAMA. 2005 May 4;293(17):2109-17. doi: 10.1001/jama.293.17.2109. PMID 15870414
- [Derived] Garg S, Sarno G, Serruys PW, Rodriguez AE, Bolognese L, Anselmi M, De Cesare N, Colangelo S, Moreno R, Gambetti S, Monti M, Bristot L, Bressers M, Garcia-Garcia HM, Parrinello G, Campo G, Valgimigli M; STRATEGY and MULTISTRATEGY Investigators. Prediction of 1-year clinical outcomes using the SYNTAX score in patients with acute ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention: a substudy of the STRATEGY (Single High-Dose Bolus Tirofiban and Sirolimus-Eluting Stent Versus Abciximab and Bare-Metal Stent in Acute Myocardial Infarction) and MULTISTRATEGY (Multicenter Evaluation of Single High-Dose Bolus Tirofiban Versus Abciximab With Sirolimus-Eluting Stent or Bare-Metal Stent in Acute Myocardial Infarction Study) trials. JACC Cardiovasc Interv. 2011 Jan;4(1):66-75. doi: 10.1016/j.jcin.2010.09.017. PMID 21251631
- [Derived] Valgimigli M, Campo G, Percoco G, Bolognese L, Vassanelli C, Colangelo S, de Cesare N, Rodriguez AE, Ferrario M, Moreno R, Piva T, Sheiban I, Pasquetto G, Prati F, Nazzaro MS, Parrinello G, Ferrari R; Multicentre Evaluation of Single High-Dose Bolus Tirofiban vs Abciximab With Sirolimus-Eluting Stent or Bare Metal Stent in Acute Myocardial Infarction Study (MULTISTRATEGY) Investigators. Comparison of angioplasty with infusion of tirofiban or abciximab and with implantation of sirolimus-eluting or uncoated stents for acute myocardial infarction: the MULTISTRATEGY randomized trial. JAMA. 2008 Apr 16;299(15):1788-99. doi: 10.1001/jama.299.15.joc80026. Epub 2008 Mar 30. PMID 18375998